CLINICAL TRIAL: NCT04331626
Title: An Exploratory Clinical Study of Low-dose Gemcitabine Combined With Nivolumab for Second-line and Higher-line Treatment of Driving Gene-negative Non-small Cell Lung Cancer
Brief Title: Low-dose Gemcitabine Combined With Nivolumab for Second-line and Above Line Treatment of NSCLC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019090507
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2019-12

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: PD - 1 antibodies; Low-dose Gemcitabine; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Low-dose Gemcitabine Combined With nivolumab (Experimental): Bristol-myers squibb (BMS) company's nivolumab injection liquid (trade name: odiwal). Recommended dosage: 3mg/kg, intravenously injected once every 2 weeks for 60 minutes. As long as clinical benefit is observed, continue treatment with this product for up to 6 courses. Gemcitabine hydrochloride injection from eli lilly. Use 50% of the recommended dose, i.e. 500mg/m2, intravenously for 30 minutes. Day 1 and day 8 administration. Depending on the patient's tolerance to gemcitabine, a reduced dose may be considered for each treatment cycle or one treatment cycle. Use for 1 year. If a Ⅲ magnitude of adverse reactions, it is necessary to permanently discontinued.
  Interventions: Drug: Gemcitabine Injectable Product

INTERVENTIONS:
Drug: Gemcitabine Injectable Product — Low dose chemotherapy drug combined with pd-1 antibody, Gemcitabine should be administered at 50% of the recommended dose, i.e. 500mg/m2, for 30 minutes by intravenous drip. Day 1 and day 8 administration.
  Other Names: nivolumab

SUMMARY:
In recent years, immunotherapy research has made great progress, especially the immunocheckpoint inhibitors represented by anti-pd-1 antibody have shown good efficacy in the treatment of malignant tumors, and some patients can achieve long-term survival. However, despite the encouraging clinical data, only a small number of people have benefited. Therefore, how to further improve the efficacy of immunotherapy and expand the benefit population has become the focus of this field.

The applicant was previously published in Oncoimmunology (2017; E1331807) pointed out in the above article: MDSC is a group of immunosuppressive cells, the number of this group of cells in the body of cancer patients is more than normal, its presence affects the proliferation, activation and function of T cells, is one of the important factors affecting the efficacy of immunocheckpoint inhibitors. Therefore, ideal drugs used in combination with immunocheckpoint inhibitors should meet the following conditions: first, they can kill or inactivate tumor cells to release tumor-specific or associated antigens; Second, MDSC and other immunosuppressive cells can be eliminated. Third, the number and function of T cells were not affected.

Gemcitabine is a synthetic antimetabolic tumor drug widely used in the treatment of locally advanced or metastatic non-small cell lung cancer. Myelosuppression is the dose - limiting toxicity of gemcitabine, which includes lymphocytopenia. Therefore, if the commonly used clinical dose gemcitabine is used in combination with pd-1 antibody, the effect of pd-1 antibody will be affected due to the reduction of lymphocytes caused by gemcitabine. Therefore, we speculated that the reduced-dose treatment of gemcitabine combined with pd-1 antibody might have synergistic anti-tumor effect on the second-line and above second-line treatment of non-small cell lung cancer with negative driver gene, and the adverse reactions were relatively mild.

This study is a phase IV, open, non-randomized, single-arm, single-center study to investigate the safety and efficacy of half-dose gemcitabine combined with pd-1 antibody in second-line and above treatment of non-small cell lung cancer patients with negative driver genes. Fifty subjects will be enrolled in this study. The primary endpoint of the study was ORR, while secondary endpoints included DCR, PFS, and OS.

DETAILED DESCRIPTION:
In recent years, immunotherapy research has made great progress, especially the immunocheckpoint inhibitors represented by anti-pd-1 antibody have shown good efficacy in the treatment of malignant tumors, and some patients can achieve long-term survival. However, despite the encouraging clinical data, only a small number of people have benefited. Therefore, how to further improve the efficacy of immunotherapy and expand the benefit population has become the focus of this field.

Conventional view holds that chemotherapeutic drugs work by directly killing tumor cells. In recent years, with the in-depth understanding of immunity, people have realized that the anti-cancer effect of chemotherapy drugs depends on the body's sound immune system, and chemotherapy drugs have been more and more recognized as an immune regulator. However, it should be noted that the combination of drugs may not achieve the desired results, or even the opposite.

The applicant was previously published in Oncoimmunology (2017; E1331807) pointed out in the above article: MDSC is a group of immunosuppressive cells, the number of this group of cells in the body of cancer patients is more than normal, its presence affects the proliferation, activation and function of T cells, is one of the important factors affecting the efficacy of immunocheckpoint inhibitors. Therefore, ideal drugs used in combination with immunocheckpoint inhibitors should meet the following conditions: first, they can kill or inactivate tumor cells to release tumor-specific or associated antigens; Second, MDSC and other immunosuppressive cells can be eliminated. Third, the number and function of T cells were not affected.

Gemcitabine is a synthetic antimetabolic tumor drug widely used in the treatment of locally advanced or metastatic non-small cell lung cancer. Myelosuppression is the dose - limiting toxicity of gemcitabine, which includes lymphocytopenia. Therefore, if the commonly used clinical dose gemcitabine is used in combination with pd-1 antibody, the effect of pd-1 antibody will be affected due to the reduction of lymphocytes caused by gemcitabine. Therefore, we speculated that the reduced-dose treatment of gemcitabine combined with pd-1 antibody might have synergistic anti-tumor effect on the second-line and above second-line treatment of non-small cell lung cancer with negative driver gene, and the adverse reactions were relatively mild.

This study is a phase IV, open, non-randomized, single-arm, single-center study to investigate the safety and efficacy of half-dose gemcitabine combined with pd-1 antibody in second-line and above treatment of non-small cell lung cancer patients with negative driver genes. Fifty subjects will be enrolled in this study. The primary endpoint of the study was objective efficiency (ORR), while secondary endpoints included disease control rate (DCR), disease-free progression (PFS), and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* the patient voluntarily participated in the study and signed the informed consent;
* advanced non-small cell lung cancer with negative driving gene confirmed by pathology has at least one measurable focus.
* in the last 6 months, chemotherapy failed;
* 18-70 years old; ECoG PS score 0-1; estimated survival time over 3 months;
* within 7 days before treatment, the main organ functions meet the following standards:

  1. blood routine examination standard (without blood transfusion within 14 days):

     A) hemoglobin (HB) ≥ 90g / L;

     B) neutrophil absolute value (ANC) ≥ 1.5 × 109 / L;

     C) platelet (PLT) ≥ 80 × 109 / L
  2. biochemical examination shall meet the following standards:

     A) TBIL ≤ 1.5 times the upper limit of normal value (ULN);

     B) ALT and AST ≤ 2.5 × ULN, if with liver metastasis, ALT and AST ≤ 5 × ULN;

     C) Cr ≤ 1.5 × ULN or CCR ≥ 60ml / min;
  3. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ the lower limit of normal value (50%).
* women of childbearing age shall agree to use contraceptive measures (such as IUD, contraceptive pill or condom) during the study and within 6 months after the end of the study; women of childbearing age shall agree to use contraceptive measures during the study and within 6 months after the end of the study (such as IUD, contraceptive pill or condom); women of childbearing age shall agree to use contraceptive measures during the study and 6 months after the end of the study if their pregnancy test is negative within 7 days before the study.

Exclusion Criteria:

* patients who have used PD-1 antibody of other companies before;
* with pleural effusion or ascites, it causes respiratory syndrome (≥ CTC AE Level 2 dyspnea);
* unresponsive toxic reactions higher than level 1 of CTC AE (4.0) caused by any previous treatment, excluding hair loss;
* patients with any serious and / or uncontrolled disease, including:

  1. patients with myocardial ischemia or myocardial infarction above grade I, arrhythmia (including QTc ≥ 480ms) and congestive heart failure ≥ grade 2 (NYHA classification);
  2. active or uncontrollable severe infection (≥ CTC AE Level 2 infection);
  3. renal failure needs hemodialysis or peritoneal dialysis;
* patients with any serious and / or uncontrolled disease, including:

  1. have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
  2. poor control of diabetes mellitus (FBG > 10mmol / L);
  3. routine urine test indicated that urine protein was ≥ + +, and 24-hour urine protein was more than 1.0 G;
  4. patients with epilepsy who need treatment;
* received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before the group;
* those who have a history of psychoactive drug abuse and are unable to quit or have mental disorders;
* participated in clinical trials of other anti-tumor drugs within four weeks;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 months
  The proportion of patients whose tumor volume reduction reaches the predetermined value and can maintain the minimum time limit is the sum of the proportion of complete and partial remission.

SECONDARY OUTCOMES:
Disease control rate | 3 years
  The percentage of patients with PR + Cr and SD after treatment in the number of evaluable cases, and the RECIST standard is at least 4 weeks.
disease free progression | 3 years
  The time from the beginning of treatment to the occurrence (in any respect) progression or (for any reason) death of the tumor.
overall survival | 3 years
  The time from the beginning of treatment to (for any reason) death. The last follow-up time is usually calculated as the time of death for the subjects who have lost the visit before death.

CONTACTS AND LOCATIONS:
Overall Officials: Zibing Wang, Doctor, Study Director — Henan Cancer Hospital

IPD SHARING:
Plan to Share IPD: No